CLINICAL TRIAL: NCT02251977
Title: The Effect of Monosialotetrahexosylganglioside (GM1) in Prevention of Oxaliplatin Induced Neurotoxicity in Colorectal Cancer Patients Who Received Oxaliplatin-based Adjuvant Chemotherapy: A Multi-center, Randomized, Placebo-controlled Trial
Brief Title: Effect of GM1 in Prevention of Oxaliplatin Induced Neurotoxicity in Stage II/III Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhong Li (Other)
Responsible Party: Sponsor-Investigator, Yuhong Li, MD Ph D, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GOXL-18
Record Dates: First submitted 2014-09-21; First posted 2014-09-29 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Colorectal Cancer; Chemotherapy-induced Neutropenia
MeSH Terms: conditions — Colorectal Neoplasms | interventions — G(M1) Ganglioside; XELOX; Leucovorin; Fluorouracil; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant Chemotherapy plus GM1 (Experimental): Patients will receive mFOLFOX6 (fluorouracil, leucovorin, and oxaliplatin) or XELOX (capecitabine and oxaliplatin) for adjuvant chemotherapy. While GM1 will be delivered to patients through the day before the initiation of chemotherapy (Day0) to the completion of chemotherapy (Day4), and the dosages of GM1 for patients who receive mFOLFOX6 or XELOX are 80mg or 120mg per day.
  Interventions: Drug: GM1; Drug: mFOLFOX6 or XELOX
- Adjuvant Chemotherapy plus placebo (Placebo Comparator): Patients will receive mFOLFOX6 (fluorouracil, leucovorin, and oxaliplatin) or XELOX (capecitabine and oxaliplatin) for adjuvant chemotherapy. While placebo will be delivered to patients through the day before the initiation of chemotherapy (Day0) to the completion of chemotherapy (Day4).
  Interventions: Drug: placebo; Drug: mFOLFOX6 or XELOX

INTERVENTIONS:
Drug: GM1 — GM1 will be delivered to patients through the day before the initiation of chemotherapy (Day0) to the completion of chemotherapy (Day4), and the dosages of GM1 for patients who receive mFOLFOX6 or XELOX are 80mg or 120mg per day.
  Other Names: monosialotetrahexosylganglioside
  Arms: Adjuvant Chemotherapy plus GM1
Drug: placebo — Placebo will be delivered to patients through the day before the initiation of chemotherapy (Day0) to the completion of chemotherapy (Day4), and the dosages of placebo for patients who receive mFOLFOX6 or XELOX are 80mg or 120mg per day.
  Arms: Adjuvant Chemotherapy plus placebo
Drug: mFOLFOX6 or XELOX — mFOLFOX6: Patients will receive mFOLFOX6 every 14 days, Oxaliplatin 85mg/m2 IV over 3 hours on Day1; Calcium Folinate IV over 2h on Day 1(Leucovorin 200mg/m2 or CF 400 mg/m2); 5-Fluorouracil 400mg/m2 IV on Day1; followed by 5-Fluorouracil 2.4g/m2 for 46 hours continuous infusion on Day1.
  XELOX: Patients will receive XELOX every 21 days, Oxaliplatin 130mg/m2 IV over 3 hours on Day1;followed by Capecitabine 1000mg/m2 oral twice daily for 14 days.
  The optimum chemotherapy regimen is at the discretion of the investigators based on the condition of each patient.
  Other Names: Oxalipaltin; Leucovorin; Calcium Folinate; 5-Fluorouracil; Capecitabine

SUMMARY:
The primary objective of this study is to assess the efficacy of monosialotetrahexosylganglioside (GM1) for preventing oxaliplatin induced neurotoxicity in colorectal cancer patients who received oxaliplatin-based adjuvant chemotherapy.

DETAILED DESCRIPTION:
Oxaliplatin is a key agent in the treatment of colorectal cancer. However, peripheral neuropathy markedly limits the use of oxaliplatin. Many drugs have been tried to decrease the development of oxaliplatin induced peripheral neurotoxicity, however, the results remain disappointing. This multi-center, randomized, placebo-controlled trial was performed to assess the efficacy of monosialotetrahexosylganglioside (GM1) for preventing oxaliplatin induced neurotoxicity in colorectal cancer patients who received oxaliplatin-based adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old, male or female
* Histologically confirmed diagnosis of colorectal adenocarcinoma with a phase II or III disease, within 2 months from radical resection, and intends to receive 6 months of adjuvant chemotherapy with mFOLOFX6 or XELOX, without adjuvant radiation indications
* No prior any level of peripheral nerve system disease
* Patients have not received any other possible neurotoxic-reaction-causing drugs (such as oxaliplatin, cisplatin and paclitaxel drugs etc)
* With the capability to accurately record the occurrence and severity of neurotoxicity by questionnaire
* With normal functions of major organs
* No contraindication to chemotherapy
* Life expectancy ≥ 3 months
* Patients have provided a signed Informed Consent Form

Exclusion Criteria:

* Patients who received radical resection, but are expected not be able to complete 6 months of adjuvant chemotherapy
* Patients who receive palliative chemotherapy
* Patients who need adjuvant or palliative radiotherapy during chemotherapy
* Be allergic to GM1
* Hereditary abnormal metabolism of glucose and lipid
* Doctors believe that patients are not suitable for receiving GM1 treatment
* With confirmed history of neurological or psychiatric disorders, including epilepsy and dementia
* With concomitant diseases that will seriously harm the patients' safety or impact the completion of the study
* Patients (male or female) have fertility possibility but not willing or not to take effective contraceptive measures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2014-09; Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
rates of grade 2 or more chronic cumulative neurotoxicity of both arms | 9 months
  measured by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0, with standardized questions regarding neurotoxic symptoms and examples of answers

SECONDARY OUTCOMES:
rates of chronic cumulative neurotoxicity of both arms | 9 months
  measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy 20
time to grade 2 or more neurotoxicity of both arms | 9 months
rates of dose reduction or withdrawal due to oxaliplatin induced neurotoxicity of both arms | 9 months
rates of acute neurotoxicity of both arms | 6 months
  measured by a numerical analog scale ranging from 0 to 10 that addressed sensitivity touching cold items, discomfort swallowing cold items, throat discomfort, and muscle cramps
rates and grades of adverse reactions of both arms | 6 months
rates of 3 year disease free survival of both arms | 3 years

OTHER OUTCOMES:
change degrees of the levels of nerve growth factor and other neurotrophic factors of both arms | 6 months
genetic polymorphisms of oxaliplatin induced severe and cumulative neurotoxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuhong Li, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wang DS, Wang ZQ, Chen G, Peng JW, Wang W, Deng YH, Wang FH, Zhang JW, Liang HL, Feng F, Xie CB, Ren C, Jin Y, Shi SM, Fan WH, Lu ZH, Ding PR, Wang F, Xu RH, Li YH. Phase III randomized, placebo-controlled, double-blind study of monosialotetrahexosylganglioside for the prevention of oxaliplatin-induced peripheral neurotoxicity in stage II/III colorectal cancer. Cancer Med. 2020 Jan;9(1):151-159. doi: 10.1002/cam4.2693. Epub 2019 Nov 13. PMID 31724334